CLINICAL TRIAL: NCT01974271
Title: IMPACT OF COMORBITIES ON HEMOGLOBIN STABILITY IN CHONIC KIDNEY DISEASE PATIENTS ON DIALYSIS TREATED WITH C.E.R.A
Brief Title: An Observational Study of Hemoglobin Stability in Chronic Kidney Disease Patients on Dialysis Treated With Mircera (Methoxy Polyethylene Glycol-epoetin Beta)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28980
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, multicenter, observational study will evaluate the impact of comorbidities on hemoglobin stability in chronic kidney disease patients on dialysis treated with Mircera (methoxy polyethylene glycol-epoetin beta). Eligible patients will be followed for 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic kidney disease patients on hemodialysis or hemodiafiltration for at least 3 months
* Previously treated with an erythropoietin stimulating agent (ESA)
* Patient for whom the investigator decided to initiate treatment with Mircera for medical reasons
* Last hemoglobin level before initiation of Mircera within the range of 10-12 g/dL

Exclusion Criteria:

* Current participation in a clinical trial on renal anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease patients on hemodialysis or hemodiafiltration for at least 3 months, previously treated with an erythropoietin stimulating agent (ESA) and for whom treatment with Mircera is indicated
Sampling Method: Probability Sample
Enrollment: 661 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a variation of Hb level of +/- 1 g/dL between the first Mircera injection and Month 6 | 6 months

SECONDARY OUTCOMES:
Percentage of patients with Hb value within the range of 10 - 12 g/dL | 6 months
Change in Hb level | from baseline to Month 6
Monthly dose of Mircera | 6 months
Safety: Incidence of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (70):
- France (70):
  - Aix-en-Provence
  - Ajaccio
  - Annonay
  - Arras
  - Auch
  - Aurillac
  - Beauvais
  - Bois-Bernard
  - Bordeaux
  - Bourg-en-Bresse
  - Bourgoin
  - Brest
  - Chamalières
  - Chaumont
  - Clermont-Ferrand
  - Colmar
  - Condom
  - Dijon
  - Dourlers
  - Épinal
  - Fleurance
  - Fourmies
  - Gap
  - Gradignan
  - Haguenau
  - La Roche-sur-Yon
  - La Tronche
  - Le Mans
  - Le Puy-en-Velay
  - Libourne
  - Lille
  - Maubeuge
  - Meaux
  - Mirande
  - Montereau
  - Nantes
  - Neuilly-sur-Seine
  - Nîmes
  - Nogaro
  - Noyal-Pontivy
  - Olivet
  - Orléans
  - Paris
  - Pessac
  - Poitiers
  - Quimper
  - Quincy-sous-Sénart
  - Rambouillet
  - Rennes
  - Rezé
  - Roubaix
  - Rouen
  - Saint-Brieuc
  - Saint-Laurent-du-Var
  - Saint-Lô
  - Saint-Marcel
  - Saint-Nazaire
  - Saint-Ouen
  - Saint-Priest-en-Jarez
  - Salouël
  - Saran
  - Stains
  - Strasbourg
  - Toulouse
  - Tourcoing
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vesoul
  - Villefranche-de-Rouergue
  - Yssingeaux